CLINICAL TRIAL: NCT03969784
Title: Microparticles in Peritoneal Carcinomatosis of Colorectal Origin
Acronym: MICROCOL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-A00688-49; 2019-08 (Other: Assistance Publique Hopitaux de Marseille)
Record Dates: First submitted 2019-05-28; First posted 2019-05-31 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- colorectal cancer patient with peritoneal carcinosis (Experimental)
  Interventions: Other: blood draw, tumoral biopsy tissus
- colorectal cancer patient without metastasis (Active Comparator)
  Interventions: Other: blood draw, tumoral biopsy tissus

INTERVENTIONS:
Other: blood draw, tumoral biopsy tissus — Patient will have specific blood draw and part of their tumoral tissu biopsied

SUMMARY:
Peritoneal carcinomatosis (PC), a tumoral tumor of the peritoneum, is a frequent metastatic localization of colorectal cancer (CRC, 13%). Long regarded as a palliative situation, its management has progressed significantly with a curative treatment based on a complete cytoreduction surgery coupled with intraperitoneal hyperthermic chemotherapy. However current screening tools, tumor markers (ACE, CA19-9, CA125) and abdominopelvic CT scan are insufficient, to diagnose CP early. A non-invasive biomarker, more sensitive and more specific than currently available tumor markers, would be a major advance in oncology. Microparticles (MPs), vesicles from extracellular membrane budding in response to cell activation or apoptosis of different cell types, have been described as implicated in tumor progression, procoagulant activity associated with cancer, and initiation of metastatic niches. A specific microparticulate (microparticulosome) signature has been reported in patients with CRC, particularly in the presence of a thromboembolic event. However, there is currently no data on PMs and their involvement in CP. In addition, CP and surgery coupled with hyperthermic intraperitoneal chemotherapy are major risk factors for thromboembolic complications. The characterization of prothrombotic PMs is therefore essential to predict such event.

The main objective of this project is to characterize the microparticulate signature of CP of colorectal origin and to compare it with that of CP without CP. The secondary objectives are to compare the microparticulate signature obtained on peripheral venous samples and intraoperative tumor samples, evaluate the evolution of the microparticulate signature between the beginning and the end of the intervention, then correlate the peripheral signature to the oncological follow-up of the patients with CP and the occurrence of a thromboembolic event.

ELIGIBILITY:
Inclusion Criteria:

* patient presenting a peritoneal carcinomatosis from colorectal cancer origin

Exclusion Criteria:

* patient presenting a peritoneal carcinomatosis from other pathologies than colorectal cancer origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-03-28 (Actual); Study Completion 2025-03-03 (Actual)

PRIMARY OUTCOMES:
percentage of microparticule | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Garrido, Study Director — Assitance Publique Hopitaux de Marseille
Locations (1):
- Timone, Marseille, France

IPD SHARING:
Plan to Share IPD: No